CLINICAL TRIAL: NCT04420832
Title: Diagnostic UltraSonography for the Choice of Treatment of Acute Achilles Tendon Rupture
Brief Title: Acute Achilles Tendon Rupture - Choice of Treatment Based on Ultrasound Findings
Acronym: DUSTAR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Katarina Nilsson Helander, Principal investigator, Sahlgrenska University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATR ultrasound study
Record Dates: First submitted 2020-05-17; First posted 2020-06-09 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Achilles Tendon Rupture; Athletic Injuries; Ultrasonography; Rupture; Acute Disease
MeSH Terms: conditions — Athletic Injuries; Rupture; Acute Disease | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical treatment (Active Comparator): Patients with a distance of 5 mm or more between tendon ends will be treated surgically and with physiotherapy
  Interventions: Procedure: Surgical treatment
- Non-surgical treatment (Other): Patients with a distance of less than 5 mm between tendon ends will be treated non-surgically and with physiotherapy
  Interventions: Other: Non-surgical treatment

INTERVENTIONS:
Procedure: Surgical treatment — Se above
  Arms: Surgical treatment
Other: Non-surgical treatment — See above
  Arms: Non-surgical treatment

SUMMARY:
Patients with acute achilles tendon rupture will go through an acute ultrasound. Based on the distance between the ends of the tendon the investigators will decide if the patient is going to be treated with or without surgery.

ELIGIBILITY:
Inclusion Criteria:

* acute achilles tendon rupture diagnosed less than 48 hours from injury
* mid-substance rupture

Exclusion Criteria:

* previous achilles tendon rupture
* lower leg disability
* diabetes mellitus
* neurovascular disease
* immunosuppression
* non-Swedish speaker

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Difference in functional outcome between patients treated surgically and non-surgically | 3 months
  The primary outcome will be a comparison of function by the heel-rise work test developed by Silbernagel et al. This is a validated test which combines both the height of each heel-rise and the number of repetitions.
Difference in functional outcome between patients treated surgically and non-surgically | 6 months
  The primary outcome will be a comparison of function by the heel-rise work test developed by Silbernagel et al. This is a validated set of tests measuring vertical jump, strength and endurance
Difference in functional outcome between patients treated surgically and non-surgically | 12 months
  The primary outcome will be a comparison of function by the heel-rise work test developed by Silbernagel et al. This is a validated set of tests measuring vertical jump, strength and endurance
Difference in functional outcome between patients treated surgically and non-surgically | 24 months
  The primary outcome will be a comparison of function by the heel-rise work test developed by Silbernagel et al. This is a validated set of tests measuring vertical jump, strength and endurance

SECONDARY OUTCOMES:
Ultrasonography (US) | 6 months
  Achilles tendon length - measured using US extended field of view
Ultrasonography (US) | 12 months
  Achilles tendon length - measured using US extended field of view
Ultrasonography (US) | 24 months
  Achilles tendon length - measured using US extended field of view
Achilles Tendon Rupture Score (ATRS) | 3 months
  Patient reported outcome measure (PROM) specific for achilles tendon rupture
Achilles Tendon Rupture Score (ATRS) | 6 months
  Patient reported outcome measure (PROM) specific for achilles tendon rupture. Minimum value 0. Maximum value 100. Higher scores mean better outcome.
Achilles Tendon Rupture Score (ATRS) | 12 months
  Patient reported outcome measure (PROM) specific for achilles tendon rupture. Minimum value 0. Maximum value 100. Higher scores mean better outcome.
Achilles Tendon Rupture Score (ATRS) | 24 months
  Patient reported outcome measure (PROM) specific for achilles tendon rupture. Minimum value 0. Maximum value 100. Higher scores mean better outcome.
Physical Activity Scale (PAS) | 3 months
  PROM to measure overall physical activity. Minimum value 1. Maximum value 6. Higher scores mean a better outcome.
Physical Activity Scale (PAS) | 6 months
  PROM to measure overall physical activity. Minimum value 1. Maximum value 6. Higher scores mean a better outcome.
Physical Activity Scale (PAS) | 12 months
  PROM to measure overall physical activity. Minimum value 1. Maximum value 6. Higher scores mean a better outcome.
Physical Activity Scale (PAS) | 24 months
  PROM to measure overall physical activity. Minimum value 1. Maximum value 6. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Nilsson Helander, MD Ass Prof., Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Department of Orthopedics, Gothenburg, Västra Götalandsregionen, Sweden

IPD SHARING:
Plan to Share IPD: Undecided